CLINICAL TRIAL: NCT02829515
Title: The National Tonsil Surgery Register in Sweden
Brief Title: Tonsil Surgery in Sweden: A National Quality Register
Acronym: NTSRS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Joacim Stalfors (Other)
Collaborators: Swedish Association of Local Authorities and Regions (Other); Sahlgrenska University Hospital (Other); Karolinska Institutet (Other); Linkoeping University (Other Government); Region Örebro County (Other)
Responsible Party: Sponsor-Investigator, Joacim Stalfors, Register Director, National Tonsil Surgery Register in Sweden
Organization: National Tonsil Surgery Register in Sweden (Other)
Other Study IDs: 1111
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Tonsillectomy; Prospective Studies; Registries; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: tonsil surgery with or without concomitant adenoidectomy — tonsillectomy, tonsillectomy with adenoidectomy, tonsillotomy, tonsillectomy with adenoidectomy

SUMMARY:
For the purpose of quality assurance, the Swedish Association for Otorhinolaryngology and Head and Neck surgery has developed several national registers concerning ear, nose and throat care. One of these is the National Tonsil Surgery Registry in Sweden (NTSRS). In NTSRS patients undergoing tonsil surgery for benign indications are included. Data regarding indication, surgical methods and techniques as well as patient reported outcomes measures are collected. The register is designed to facilitate description of clinical activities in a unit and help identify the need of clinical improvement programs. By compiling national data, the register can be used to describe clinical practice in a large national cohort.

DETAILED DESCRIPTION:
The National Tonsil Surgery Register in Sweden (NTSRS), started in 1997 as one among several registers, aimed to reinforce quality in the Swedish health care and were revised 2009. Data in the NTSRS are collected through four questionnaires; two are filled in by the ENT-surgeon and two postoperative forms, filled in by the patient or the legal guardian, collecting patient related outcome measures (PROM) 30 respective 180 days after surgery.

In the first surgeon questionnaire age, sex, social security number and indication for surgery (upper airway obstruction, recurrent tonsillitis, chronic tonsillitis, peritonsillar abscess, and systemic complications because of tonsillitis or other) are recorded. This is filled in when surgery is notified.

The second surgeon questionnaire records surgical method (TE, TEA, TT or TTA), surgical instruments used for dissection (cold steel, radiofrequency, diathermy scissors, ultracision or other) and hemostasis method used (injection with epinephrine, unipolar diathermy, bipolar diathermy, ties, suture ligature, radiofrequency, other or "none other than compression with packs"). The questionnaire also records information regarding daycare/inpatient procedure and primary postoperative bleeding. Due to the configuration of the questionnaires and the ambition to cover both inpatient and daycare procedures, primary bleeding is defined as bleeding during hospitalization.

The first patient/caregiver form contains several questions mainly regarding postoperative complications. Any contact with healthcare provider due to postoperative bleeding/pain/infection as well as consequences of the contact; prescribed antibiotics and readmission/return to theatre are reported. Conformity between preoperative information and actual patient experience was is also included in this form.

The final questionnaire that is sent to the second patient/caregiver questionnaire asks for perceived symptom relief after 180 days by choosing one alternative of four statements: My symptoms are gone / My symptoms are almost gone / My symptoms have not disappeared/ My symptoms have worsened.

In order to assess coverage for the NTSRS, data has been matched on an individual level with another national register, the National Patient Register (NPR). The NPR is managed by the National Board of Health and Welfare and registration of surgical procedures is mandatory by law for all physicians in Sweden. The coverage of NTSRS for the study period 2012-2014 was 75%, 81.4% and 80.7% respectively

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing benign tonsil surgery in Sweden

Exclusion Criteria:

* All patients operated with an C- or D0-48 ICD 10 code, indicating not benign diagnoses

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing benign tonsil surgery in Sweden
Sampling Method: Non-Probability Sample
Enrollment: 11000 (Estimated)
Dates: Start 2009-05 (Actual); Primary Completion 2012-03-01 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Patient reported symptom relief | 6 months postoperative report
  The final questionnaire that is sent to the second patient/caregiver questionnaire asks for perceived symptom relief after 180 days by choosing one alternative of four statements: My symptoms are gone / My symptoms are almost gone / My symptoms have not disappeared/ My symptoms have worsened.

SECONDARY OUTCOMES:
Patient reported postoperative bleeding | 30 days postoperative report
  The first patient/caregiver form contains several questions mainly regarding postoperative complications. Any contact with healthcare provider due to postoperative bleeding/pain/infection as well as consequences of the contact; prescribed antibiotics and readmission/return to theatre are reported. Conformity between preoperative information and actual patient experience was is also included in this form.

CONTACTS AND LOCATIONS:
Overall Officials: Joacim Stalfors, MD, PhD, Study Director — Sahlgrenska Academy
Locations (1):
- National Tonsil Surgery Register in Sweden, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All registered data i available online for registrating units.
URL: https://ton.registercentrum.se/

REFERENCES:
- [Background] Odhagen E, Sunnergren O, Hemlin C, Hessen Soderman AC, Ericsson E, Stalfors J. Risk of reoperation after tonsillotomy versus tonsillectomy: a population-based cohort study. Eur Arch Otorhinolaryngol. 2016 Oct;273(10):3263-8. doi: 10.1007/s00405-015-3871-7. Epub 2016 Jan 4. PMID 26728487
- [Background] Gerhardsson H, Stalfors J, Odhagen E, Sunnergren O. Pediatric adenoid surgery in Sweden 2004-2013: Incidence, indications and concomitant surgical procedures. Int J Pediatr Otorhinolaryngol. 2016 Aug;87:61-6. doi: 10.1016/j.ijporl.2016.05.020. Epub 2016 May 20. PMID 27368444
- [Background] Ostvoll E, Sunnergren O, Ericsson E, Hemlin C, Hultcrantz E, Odhagen E, Stalfors J. Mortality after tonsil surgery, a population study, covering eight years and 82,527 operations in Sweden. Eur Arch Otorhinolaryngol. 2015 Mar;272(3):737-43. doi: 10.1007/s00405-014-3312-z. Epub 2014 Oct 2. PMID 25274044
- [Background] Ostvoll E, Sunnergren O, Stalfors J. Increasing Readmission Rates for Hemorrhage after Tonsil Surgery: A Longitudinal (26 Years) National Study. Otolaryngol Head Neck Surg. 2018 Jan;158(1):167-176. doi: 10.1177/0194599817725680. Epub 2017 Aug 22. PMID 28828912
- [Background] Sunnergren O, Odhagen E, Stalfors J. Incidence of second surgery following pediatric adenotonsillar surgery: a population-based cohort study. Eur Arch Otorhinolaryngol. 2017 Jul;274(7):2945-2951. doi: 10.1007/s00405-017-4543-6. Epub 2017 Mar 23. PMID 28337533
- [Background] Borgstrom A, Nerfeldt P, Friberg D, Sunnergren O, Stalfors J. Trends and changes in paediatric tonsil surgery in Sweden 1987-2013: a population-based cohort study. BMJ Open. 2017 Jan 13;7(1):e013346. doi: 10.1136/bmjopen-2016-013346. PMID 28087550
- [Result] Elinder K, Soderman AC, Stalfors J, Knutsson J. Factors influencing morbidity after paediatric tonsillectomy: a study of 18,712 patients in the National Tonsil Surgery Register in Sweden. Eur Arch Otorhinolaryngol. 2016 Aug;273(8):2249-56. doi: 10.1007/s00405-016-4001-x. Epub 2016 Mar 28. PMID 27020269
- [Result] Soderman AC, Odhagen E, Ericsson E, Hemlin C, Hultcrantz E, Sunnergren O, Stalfors J. Post-tonsillectomy haemorrhage rates are related to technique for dissection and for haemostasis. An analysis of 15734 patients in the National Tonsil Surgery Register in Sweden. Clin Otolaryngol. 2015 Jun;40(3):248-54. doi: 10.1111/coa.12361. PMID 25515059
- [Result] Sunnergren O, Hemlin C, Ericsson E, Hessen-Soderman AC, Hultcrantz E, Odhagen E, Stalfors J. Radiofrequency tonsillotomy in Sweden 2009-2012. Eur Arch Otorhinolaryngol. 2014 Jun;271(6):1823-7. doi: 10.1007/s00405-013-2867-4. Epub 2013 Dec 24. PMID 24366615
- [Result] Hultcrantz E, Ericsson E, Hemlin C, Hessen-Soderman AC, Roos K, Sunnergren O, Stalfors J. Paradigm shift in Sweden from tonsillectomy to tonsillotomy for children with upper airway obstructive symptoms due to tonsillar hypertrophy. Eur Arch Otorhinolaryngol. 2013 Sep;270(9):2531-6. doi: 10.1007/s00405-013-2374-7. Epub 2013 Feb 6. PMID 23385384
- [Result] Stalfors J, Ericsson E, Hemlin C, Hultcrantz E, Mansson I, Roos K, Hessen Soderman AC. Tonsil surgery efficiently relieves symptoms: analysis of 54 696 patients in the National Tonsil Surgery Register in Sweden. Acta Otolaryngol. 2012 May;132(5):533-9. doi: 10.3109/00016489.2011.644252. Epub 2012 Jan 11. PMID 22235871
- [Result] Hessen Soderman AC, Ericsson E, Hemlin C, Hultcrantz E, Mansson I, Roos K, Stalfors J. Reduced risk of primary postoperative hemorrhage after tonsil surgery in Sweden: results from the National Tonsil Surgery Register in Sweden covering more than 10 years and 54,696 operations. Laryngoscope. 2011 Nov;121(11):2322-6. doi: 10.1002/lary.22179. Epub 2011 Oct 12. PMID 21994191
- [Result] Odhagen E, Sunnergren O, Soderman AH, Thor J, Stalfors J. Reducing post-tonsillectomy haemorrhage rates through a quality improvement project using a Swedish National quality register: a case study. Eur Arch Otorhinolaryngol. 2018 Jun;275(6):1631-1639. doi: 10.1007/s00405-018-4942-3. Epub 2018 Mar 24. PMID 29574597
- [Result] Alm F, Stalfors J, Nerfeldt P, Ericsson E. Patient reported pain-related outcome measures after tonsil surgery: an analysis of 32,225 children from the National Tonsil Surgery Register in Sweden 2009-2016. Eur Arch Otorhinolaryngol. 2017 Oct;274(10):3711-3722. doi: 10.1007/s00405-017-4679-4. Epub 2017 Aug 16. PMID 28815308
- [Result] Hallenstal N, Sunnergren O, Ericsson E, Hemlin C, Hessen Soderman AC, Nerfeldt P, Odhagen E, Ryding M, Stalfors J. Tonsil surgery in Sweden 2013-2015. Indications, surgical methods and patient-reported outcomes from the National Tonsil Surgery Register. Acta Otolaryngol. 2017 Oct;137(10):1096-1103. doi: 10.1080/00016489.2017.1327122. Epub 2017 Jun 9. PMID 28598766
- [Result] Gudnadottir G, Tennvall GR, Stalfors J, Hellgren J. Indirect costs related to caregivers' absence from work after paediatric tonsil surgery. Eur Arch Otorhinolaryngol. 2017 Jun;274(6):2629-2636. doi: 10.1007/s00405-017-4526-7. Epub 2017 Mar 14. PMID 28289832